CLINICAL TRIAL: NCT05893602
Title: Systemic Metal Ion Concentrations in Patients With a PEEK HD Coupling Mechanism in Modular Mega-prostheses of the Knee; a Prospective Cohort Pilot Study
Brief Title: Metal-ions in Patients With the PEEK HD Coupling Mechanism of the Knee
Acronym: MIONS
Status: Not yet recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Michiel AJ van de sande, MD, PhD, Michiel AJ van de Sande, MD, PhD, Leiden University Medical Center
Other Study IDs: NL82185.058.22
Record Dates: First submitted 2023-04-21; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Mutars; Modular Universal Tumor And Revision System; Metal-ions; Tumor Prosthesis; Megaprosthesis; PEEK-HD Coupling Mechanism; Knee Endoprosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary tumor prosthesis of the knee containing the PEEK HD coupling mechanism: This group consists of patients with a primary MUTARS knee endoprosthesis containing the PEEK-HD coupling mechanism.
  Interventions: Other: Blood sample analysis
- Revision tumor prosthesis of the knee containing the PEEK-HD coupling mechanism: This group consists of patients requiring revision surgery of their MUTARS knee endoprosthesis containing the MoM coupling mechanism (for any reason), which is exchanged/revised for the PEEK-HD coupling mechanism.
  Interventions: Other: Blood sample analysis

INTERVENTIONS:
Other: Blood sample analysis — Blood sample analysis on Cobalt and Chrome will be performed during the period under study.

SUMMARY:
The goal of this observational study is to evaluate the changes of serum metal ion (Cobalt and Chrome) levels at 0, 3-6, 12, and 24 months postoperative in patients receiving a MUTARS mega-prostheses of the knee with a PEEK HD coupling mechanism. The main question(s) to answer are: • [what is the change in serum level metal ions (Cobalt and Chrome) in patients receiving a primary MUTARS knee endoprosthesis with the PEEK HD coupling mechanism ] • [what is the change in serum level metal ions (Cobalt and Chrome) in patients with a MoM coupling mechanism revised to the PEEK HD coupling mechanism]. Participants will be asked to fill out functional outcome measures during the period under study.

DETAILED DESCRIPTION:
Rationale:

Local release of metal ions and their systemic sequelae is an increasing source of concern in patients with an endoprosthetic reconstruction of major joints. It is assumed that metal-on-metal (MoM) articulations, used in several types of mega-prostheses, may cause release of metal ions. Corrosion of non-articulating surfaces, abrasive wear of soft tissues and fretting of modular junctions could contribute to this release. The release of metal ions are known to induce inflammatory responses and immune reactions in the directly exposed tissues and can cause serious local adverse reactions such as metallosis, osteolysis, pseudotumor formation and systemic adverse effects such as cardiovascular and neurological adverse effects. Our study group previously found significantly elevated serum levels of Silver (Ag), Chrome (Cr) and Cobalt (Co) in a series (not published yet) of 11 patients with a MoM coupling mechanism of knee endoprostheses. Furthermore, a number of early mechanical failures of these MoM coupling mechanisms were encountered by the investigators recently.

The implant manufacturer (ImplantCast GmbH) recently introduced a carbon-reinforced PEEK HD (polyether ether ketone high demand) coupling mechanism in an attempt to reduce the risk of early mechanical failure and to lower the risk on the release of metal ions. Based on the outcomes of previous research and the mechanical failures of the MoM coupling mechanism, the investigating center will switch to the use of the new (approved and CE-marked) PEEK HD coupling mechanism. Hypothesized is that the PEEK HD coupling mechanism will not result in elevated serum metal ion levels in patients receiving a mega prosthesis.

Objective:

The aim is to 1) monitor and investigate the change in serum metal ion (Cobalt and Chrome) levels postoperatively (at 0, 3-6, 12 and 24 months) in patients receiving a primary PEEK HD coupling mechanism, monitor and investigate the change in serum metal ion levels pre-and postoperatively in patients with an MoM coupling mechanism which is revised to a PEEK HD coupling mechanism (in case of failure for any reason), 2) document adverse effects caused by metal ions, 3) report factors (possibly) correlating with metal ion release and 4) evaluate the functional outcome of the patient using the Patient-Reported Outcome Measurement Information System (PROMIS) 29 and or Toronto Extremity Salvage Score (TESS) lower extremity.

Study design:

This is a prospective cohort pilot study to evaluate metal ion concentrations, possible adverse effects and functional outcomes after the implantation of a PEEK HD coupling mechanism.

Study population:

Patients ≥18 years receiving a reconstruction with a MUTARS knee endoprosthesis (distal femur, proximal tibia or total knee) with a PEEK HD couplingmechanism, and patients receiving a PEEK HD coupling mechanism in the case of a revision procedure of a MUTARS knee endoprosthesis with a MoM coupling mechanism.

Main study parameters/endpoints:

(1) Serum metal ion concentrations Cobalt (Co) and Chrome (Cr) pre- and postoperatively (at 3-6, 12 and 24 months), (2) Secondary parameters are used to identify any adverse effects in patients with increased serum levels of ion metals (metallosis, osteolysis, periprosthetic loosening, pseudotumor formation). (3) Tertiary parameters are used to identify possible risk factors correlating with metal-ion release. (4) quaternary parameters (PROMIS 29 or TESS) are used to evaluate the functional outcome of the patient. All other variables (e.g. general baseline characteristics, treatment characteristics, and surgical details including prosthesis details) will be gathered within the "MORE" cohort study and "biobank" study (study number 2022-031, reference BWD005/SH/sh).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Serum metal ion concentrations (Cobalt and Chrome) will be determined at 0, 3-6, 12, and 24 months postoperatively. The potential benefits of routine determination of metal ion concentrations are early detection of toxic values of metal ions. Except for the negligible risks of routine venepuncture no potential risks are anticipated.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria: The patient

1. is 18 years of age or older
2. receives a MUTARS knee replacement with PEEK HD coupling mechanism, or undergoes a revision (for any reason) of a MUTARS knee replacement during which the MoM coupling mechanism is revised for a PEEK HD coupling mechanism
3. Is able to give informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Anamnestic use of metal containing nutritional supplements or medications
2. Contact with metal ions in the work environment
3. Renal insufficiency defined as an eGFR<60
4. Presence of implants containing Cobalt and Chrome (including non-orthopaedic implants such as stents and dental implants)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be drawn from the outpatient clinic of the orthopaedic surgery in the Leiden University Medical Center (LUMC). Starting from January 2023, all patients with an indication for a mega-prosthesis of the knee, will receive a PEEK HD coupling mechanism primarily or in case of a revision procedure (if clinically possible) after replacing the MoM coupling mechanism. Patients will be screened for eligibility by the orthopaedic surgeon. After the patient is deemed eligible, he/she will be informed about this study and asked for participation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum metal ion levels (Cobalt and Chrome) | 24 months
  Main study parameter are the change in serum metal ion levels (Cobalt/Chrome) in patients receiving the PEEK HD coupling mechanism in a MUTARS knee mega prosthesis.
  Serum metal ion levels will be obtained postoperative (at 3-6, 12 and 24 months) of patients receiving a primary MUTARS knee mega prosthesis with the PEEK HD coupling mechanism. Furthermore, serum metal ion levels will be determined pre- and postoperatively (0, 3-6, 12 and 24 months) in patients requiring revision surgery of the MoM coupling mechanism (for any reason) which is exchanged for the PEEK HD coupling mechanism.

SECONDARY OUTCOMES:
Adverse effects | 24 months
  Secondary endpoint is the emergence of adverse effects. No solid evidence for expected adverse effects is available. Therefore patients will be screened for local and systemic adverse events. No invasive examinations for low incidence adverse effects will be performed. X-rays will be performed according to standard care and are assessed for mechanical failure, osteolysis and loosening. Depending on the indication for the primary procedure (e.g. tumor type), additional imaging will be performed according to standard follow-up protocols. In case of a malignant bone tumor, magnetic resonance imaging (MRI) will be performed at one and two year follow-up to assess (pseudo)tumor formation/recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands